CLINICAL TRIAL: NCT02698202
Title: Randomized Controlled Trial to Evaluate the Efficacy of Digital Breast Tomosynthesis in Reggio Emilia Breast Cancer Screening Program in the 45-74 Age Group
Brief Title: Screening for Breast Cancer With Digital Breast Tomosynthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: Regione Emilia-Romagna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Screening
Other Study IDs: ReTomo
Record Dates: First submitted 2016-02-26; First posted 2016-03-03 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Tomosynthesis,sensitivity,specificity,screening,mammography
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Digital Breast Tomosynthesis (Experimental): to the experimental arm will be offered twice screening examination: standard 2D mammography + Digital Breast Tomosynthesis
  Interventions: Device: Digital Breast Tomosynthesis
- standard mammography (No Intervention): to the control arm the usual 2D standard mammography exam will be offered

INTERVENTIONS:
Device: Digital Breast Tomosynthesis — twice screening examination: standard 2D mammography + Digital Breast Tomosynthesis
  Arms: Digital Breast Tomosynthesis

SUMMARY:
Randomized trial comparing the performance of tomosynthesis and 2D Digital Mammography vs 2D Digital Mammography only in respect to incidence of advanced cancers (interval and following round) and interval cancers.

DETAILED DESCRIPTION:
The investigators conduct a randomized trial (about 20000 tests in the intervention arm) comparing the performance of tomosynthesis plus 2D Digital Mammography vs usual care (2D digital mammography) in respect to incidence of advanced cancers (interval and following round) and interval cancers. The investigators also will measure detection rates, specificity, interval cancers, advanced cancers occurring as interval cancers or at subsequent screens and allowing to estimate overdiagnosis. In Reggio Emilia a population-based screening program is active. It invites all women from 45 to 74 years old for a 2D digital mammography (2 projections, double reading) every 2 years (annually from 45 to 49).

Women will be asked for informed consent when they attend the mammography. I they accept they will be randomised to one of the two arms.

All examinations will be read by two independent radiologists, in case of discordance a third reading is asked.

ELIGIBILITY:
Inclusion Criteria:

45-70 years old women invited to breast cancer screening program who accepted to participate

Exclusion Criteria:

* previous breast cancer diagnosis
* pregnancy or suspicion of pregnancy
* presence of BRCA1/2 gene mutation
* Previous Digital Breast Tomosynthesis performed
* unable to understand informed consent
* chemotherapy in progress
* presence of breast implant

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26877 (Actual)
Dates: Start 2014-03-10 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of T2+ cancers after screening | 2 years
incidence of interval cancers | 2 years

SECONDARY OUTCOMES:
Detection rate | 2 years
recall rate | baseline
Positive Predictive value | baseline
diagnostic agreement between tomosynthesis and 2d mammography | baseline
Detection rate of in situ ductal carcinoma | 2 years
biopsy rate | baseline
self-reported pain and discomfort during mammography | baseline
x-ray dose | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Pattacini, MD, Principal Investigator — Inter-Institutional Imaging Department, IRCCS-Arcispedale Santa Maria Nuova, Viale Umberto I 50, 42123, Reggio Emilia, Italy
Locations (1):
- Azienda Sanitaria Locale Reggio Emilia, Reggio Emilia, Italy

REFERENCES:
- [Derived] Pattacini P, Nitrosi A, Giorgi Rossi P, Duffy SW, Iotti V, Ginocchi V, Ravaioli S, Vacondio R, Mancuso P, Ragazzi M, Campari C; RETomo Working Group. A Randomized Trial Comparing Breast Cancer Incidence and Interval Cancers after Tomosynthesis Plus Mammography versus Mammography Alone. Radiology. 2022 May;303(2):256-266. doi: 10.1148/radiol.211132. Epub 2022 Feb 1. PMID 35103537